CLINICAL TRIAL: NCT05136053
Title: A Phase 1, 3-Part, Single Ascending Dose, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Lu AG22515 (APB-A1) in Healthy Adult Subjects
Brief Title: A Study Investigating Lu AG22515 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 20119A; APB-A1-101 (Other: AprilBio Co.); NCT05303246 (obsolete NCT alias)
Record Dates: First submitted 2021-10-13; First posted 2021-11-26 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A: Lu AG22515 (Experimental): Participants will receive a single intravenous (IV) infusion of Lu AG22515.
  Interventions: Drug: Lu AG22515
- Part A: Placebo (Placebo Comparator): Participants will receive a single IV infusion of placebo matching to Lu AG22515.
  Interventions: Drug: Placebo
- Part B: Lu AG22515 and Immune System Activator (Experimental): Participants will receive a single IV infusion of Lu AG22515 and a subcutaneous (SC) injection of immune system activator 14 days prior to and 14 days following the start of Lu AG22515 IV infusion.
  Interventions: Drug: Lu AG22515; Drug: Immune System Activator
- Part B: Placebo and Immune System Activator (Placebo Comparator): Participants will receive a single IV infusion of placebo matching to Lu AG22515 and an SC injection of immune system activator 14 days prior to and 14 days following the start of placebo IV infusion.
  Interventions: Drug: Placebo; Drug: Immune System Activator
- Part C: Lu AG22515 (Experimental): Participants will receive a single intravenous (IV) infusion of Lu AG22515.
  Interventions: Drug: Lu AG22515
- Part C: Placebo (Placebo Comparator): Participants will receive a single IV infusion of placebo matching to Lu AG22515.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lu AG22515 — sterile solution for infusion
  Other Names: APB-A1
  Arms: Part A: Lu AG22515; Part B: Lu AG22515 and Immune System Activator; Part C: Lu AG22515
Drug: Placebo — sterile solution for infusion
  Arms: Part A: Placebo; Part B: Placebo and Immune System Activator; Part C: Placebo
Drug: Immune System Activator — sterile powder for injection
  Arms: Part B: Lu AG22515 and Immune System Activator; Part B: Placebo and Immune System Activator

SUMMARY:
The main goal of this study is to learn more about the safety of a drug called Lu AG22515. During the trial, healthy adult participants will receive a single dose of Lu AG22515 or a placebo (normal saline solution).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥18.0 and ≤32.0 kilograms (kg)/square meter (m^2) and weight between 55 and 110 kg (both inclusive) at screening.
* Fully vaccinated against COVID-19, as evidenced by presentation of a vaccine card. The last administration of the COVID-19 vaccination must be received a minimum of 30 days and maximum 6 month prior to dosing in this study.
* Medically healthy with no clinically significant medical history, physical examination and neurological assessment, laboratory profiles, vital signs, or electrocardiograms (ECGs), as deemed by the principal investigator (PI) or designee.

Part C only:

* The participant is Japanese, defined as being born in Japan and having four Japanese grandparents as well as living a Japanese lifestyle as confirmed by the Japanese lifestyle questionnaire.

Exclusion Criteria:

* Reported history of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
* Received any vaccination in the last 30 days prior to Day 1.

Note: Other inclusion and exclusion criteria may apply.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-08-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | From the day of study drug administration (Day 1) up to end of study (Day 113)

SECONDARY OUTCOMES:
Number of Participants With Anti-Drug Antibodies (ADAs) | Day 1 (within 2 hours prior to the start of infusion) up to end of study (Day 113)
Area Under the Concentration-Time Curve From Time 0 to Extrapolated to Infinity (AUC0-inf) of Lu AG22515 | Day 1 (within 2 hours prior to the start of infusion) up to end of study (Day 113)
Maximum Observed Plasma Concentration (Cmax) of Lu AG22515 | Day 1 (within 2 hours prior to the start of infusion) up to end of study (Day 113)
Time to Reach Cmax (Tmax) of Lu AG22515 | Day 1 (within 2 hours prior to the start of infusion) up to end of study (Day 113)
Apparent Elimination Half-life (t1/2) of Lu AG22515 | Day 1 (within 2 hours prior to the start of infusion) up to end of study (Day 113)
Apparent Total Serum Clearance (CL) of Lu AG22515 | Day 1 (within 2 hours prior to the start of infusion) up to end of study (Day 113)
Volume of Distribution During the Terminal Elimination Phase (Vz) After IV Administration of Lu AG22515 | Day 1 (within 2 hours prior to the start of infusion) up to end of study (Day 113)
Mean Residence Time (MRT) of Lu AG22515 | Day 1 (within 2 hours prior to the start of infusion) up to end of study (Day 113)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — H. Lundbeck A/S
Locations (2):
- United States (2):
  - CenExel CNS, Long Beach, California
  - Frontage Clinical Research Inc, Secaucus, New Jersey